CLINICAL TRIAL: NCT07379060
Title: Pilot Study to Evaluate a Non-invasive Training System for Inspiratory Muscles in Athletic Women
Brief Title: Non-invasive Training of the Inspiratory Muscles in Athletic Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Rocío Abalo, Principal investigator, University of Vigo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CEIm 2562
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Muscles

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Training routine and additionally perform Inspiratory Muscle Training 1 (Experimental): The experimental 1 group will follow their regular training routine and additionally perform Inspiratory Muscle Training using the PwB Medic Plus device. This training consists of 30 breaths, twice daily, with a resistance load set between 40% and 60% of their Maximum Inspiratory Pressure. The intervention will last for 10 weeks
  Interventions: Device: Inspiratory Muscle Training 1
- Training routine and additionally perform Inspiratory Muscle Training 2 (Experimental): The experimental 2 group will follow their regular training routine and additionally perform Inspiratory Muscle Training using the PwB Medic Plus device. This training consists of 30 breaths, twice daily, with a resistance load set between 40% and 60% of their Maximum Inspiratory Pressure. The intervention will last for 10 weeks
  Interventions: Device: Inspiratory Muscle Training 2
- Normal Training routine 1 (No Intervention): Normal Training routine 1
- Normal Training routine 2 (No Intervention): Normal Training routine 2

INTERVENTIONS:
Device: Inspiratory Muscle Training 1 — Inspiratory Muscle Training using the no invasive device. This training consists of 30 breaths, twice daily, with a resistance load set between 40% and 60% of their Maximum Inspiratory Pressure. The intervention will last for 10 weeks
  Arms: Training routine and additionally perform Inspiratory Muscle Training 1
Device: Inspiratory Muscle Training 2 — Inspiratory Muscle Training using the no invasive device. This training consists of 30 breaths, twice daily, with a resistance load set between 40% and 60% of their Maximum Inspiratory Pressure. The intervention will last for 10 weeks
  Arms: Training routine and additionally perform Inspiratory Muscle Training 2

SUMMARY:
The goal of this clinical trial is to study whether there are significant differences between the control and experimental groups in terms of the improvement in lung function of the athletes who have performed Inspiratory muscle training with powerbreath. The main question it aims to answer is:

• the study that power breath is effective in providing improvements in inspiratory muscle strength, lung function, exercise capacity, quality of life, analytical parameters, dyspnea, fatigue and activities of daily living and impacting their sporting success.

Researchers will compare specific powerbreath training with nettraining period without this device.

Participants will:

* Perform regular sports training along with powerbreath training for 10 weeks
* A washout period of two months
* Perform regular sports training for 10 weeks

ELIGIBILITY:
Inclusion Criteria:

* Female athletes from the Galician Center for Sports Technification (CGTD) in the city of Pontevedra.
* Sign the informed consent document.
* Possession of the mental capacity required to participate in the study

Exclusion Criteria:

* Age below the legal healthcare age (16 years).
* Lack of skills necessary to operate the no invasive device

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Power breath. Maximum Inspiratory Pressure | From enrollment to the end of treatment at 10 weeks
  This training consists of 30 breaths, twice daily, with a resistance load set between 40% and 60% of their Maximum Inspiratory Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy, Pontevedra, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No